CLINICAL TRIAL: NCT05527262
Title: Is Intensive Upper Limb Rehabilitation Effective in Chronic Stroke Patients? A Randomised Controlled Trial
Brief Title: Intensive Upper Limb Training in Chronic Stroke
Acronym: INTENSIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TBC
Record Dates: First submitted 2022-06-29; First posted 2022-09-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: upper limb; intensive training; motor impairment; kinematics; neurophysiology
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Queen Square Upper limb training programme (Experimental): Patients will undergo 45-60 hours of conventional physiotherapy and occupational therapy over 3 weeks as part of the Queen Square Upper Limb Neurorehabilitation Programme (QSUL) (Ward et al., 2019).
  Interventions: Behavioral: Queen Square Upper Limb Neurorehabilitation Programme
- Mindpod Dolphin (Experimental): Patients will undergo 45-60 hours of arm, hand and finger training using immersive gaming technology (e.g. MindPod Dolphin) over 3 weeks.
  Interventions: Device: Immersive gaming therapy
- Wait-list Control (No Intervention): Patients will receive no planned treatment but will be on a waiting list for QSUL Programme after their follow up period if over.

INTERVENTIONS:
Behavioral: Queen Square Upper Limb Neurorehabilitation Programme — A timetable will be implemented including a minimum of 45 hours of active time on task over 3 weeks 5-days a week (first and last day will involve the assessment procedures) (timetabled, 90-hours). Our unpublished in-service audits suggest that this equates to 45-60 hours of active upper limb training. The remainder of the time is spent on rest (in-session, between-session), cardiovascular fitness, and education (promoting self-efficacy). The programme is staffed with a 1:1 staff/patient ratio (4 physiotherapists, 4 occupational therapists, 4 rehabilitation assistants for 12 patients at any one time). Participants in this trial will receive two daily sessions each of physiotherapy and occupational therapy, supplemented with tailored, individualised interventions delivered by rehabilitation assistants either singly or in groups.
  Arms: Queen Square Upper limb training programme
Device: Immersive gaming therapy — The treatment group will receive a minimum of 45 hours of active time on task over 3 weeks, 5 days a week (first and last day will involve the assessment procedures) to complete arm, hand and finger training (overseen by a physiotherapist). Patients will engage with MindPod Dolphin (shoulder/elbow) and other interfaces (hand/fingers) in a customised immersive game-based platform set.
  Arms: Mindpod Dolphin

SUMMARY:
The evidence supporting routine provision of high-dose, high-intensity upper limb neurorehabilitation treatment for stroke survivors beyond the first few months after stroke is limited. The Queen Square Upper Limb (QSUL) programme provides 90 hours of upper limb neurorehabilitation over 3-weeks to chronic stroke survivors. The recently published service evaluation demonstrated encouragingly large, clinically meaningful effects at the level of activity and body function. An alternative way to deliver high doses of effective therapy is through technological developments, e.g. immersive interactive gaming environments such as the MindPod Dolphin programme.

The intention of this study is to provide stronger level evidence for intensive upper limb rehabilitation by conducting a randomised controlled trial of two different types of upper limb training compared to usual care. Patients considered suitable for the QSUL programme will be randomised to either: Group 1- intensive upper limb rehabilitation programme (QSUL); Group 2- MindPod programme; Group 3-wait-list control (who will be offered the treatment after the waiting list is complete).

The first aim of the study is to compare the effect of each type of high-dose, high-intensity upper limb training to usual care using measures of upper limb impairment and activity levels 3 months after treatment is complete.

The secondary aims are to comply with recent recommended by the Stroke Recovery and Rehabilitation Roundtable, and (i) investigate the effects of upper limb neurorehabilitation on kinematics of upper limb movement (using a KINARM exoskeleton), and (ii) use neuroimaging (MRI and EEG) and neurophysiological (TMS) measures to determine the characteristics of stroke survivors who are most likely to benefit from this treatment approach.

The results from this work will (i) help determine the impact of two methods of high dose, high intensity upper limb training in chronic stroke patients; (ii) identify whether there are any predictors of treatment response that will help stratify patients in future clinical trials of upper limb neurorehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. A first-ever unilateral stroke (ischaemic or haemorrhagic) as defined by WHO at least 6-months previously;
2. Moderate upper limb impairment as defined by Fugl-Meyer Upper Extremity (Woodbury et al., 2013) score between 19-46 (to avoid ceiling and floor effects);
3. Must be able to voluntarily extend the thumb and/or 2 or more fingers of the affected hand (10° or more)

Exclusion Criteria:

1. Other neurological diagnoses;
2. Serious communication, cognitive and language deficits (<7 on shortened version Montreal Cognitive Assessment or < 34 on Cognitive assessment scale for stroke patients);
3. Post-stroke frozen shoulder;
4. Increased muscle tone in wrist/finger extensors (≥3 on Modified Ashworth Scale);
5. Loss of passive range in any upper limb joints;
6. Fatigue of <30 on the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale;
7. Apraxia score of <5 on the TULIA assessment;
8. Severe shoulder pain measured by Chedoke Impairment Inventory: Stage of Shoulder Pain 1, 2, and 3;
9. Vision impairment that impedes seeing the television screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Upper Extremity Assessment | Three-months follow-up
  Upper limb motor impairment measure, with a minimum score of 0 and a maximum score of 60 (excluding reflexes, Woodbury et al., 2007). A higher score means a better upper limb motor impairment outcome.

SECONDARY OUTCOMES:
Fugl Meyer Upper Extremity Assessment | Baseline and 3 weeks post-intervention
  Upper limb motor impairment measure, with a minimum score of 0 and a maximum score of 60 (excluding reflexes, Woodbury et al., 2007). A higher score means a better upper limb motor impairment outcome.
Action Research Arm Test | Baseline, 3 weeks post-intervention and three-months follow-up
  Upper limb function and dexterity measure with a minimum score of 0 and a maximum score of 57. A higher score means a better upper limb function and dexterity outcome.
Chedoke Arm and Hand Activity Inventory (CAHAI-13) | Baseline, 3 weeks post-intervention and three-months follow-up
  Upper limb function measure with a minimum score of 13 and maximum score of 91. A higher score indicating a better upper limb function outcome.
Stroke Impact Scale | Baseline, 3 weeks post-intervention and three-months follow-up
  Disability and quality of life measure with a minimum score of 0 and a maximum score of 100. A higher score indicating a higher quality of life.
Quality of life (EQ-5D5L) | Baseline, 3 weeks post-intervention and three-months follow-up
  Quality of Life measure with a minimum score of 1,1,1,1,5 and a maximum score of 5,5,5,5,5. A higher score means more severe and frequent problems.
The stroke self-efficacy questionnaire | Baseline, 3 weeks post-intervention and three-months follow-up
  Self-efficacy measure involving 3-item self-report scale measuring self-efficacy judge- ments in specific domains of functioning post stroke. Individuals rate their belief in their ability to achieve each of the 13 items on a 10-point scale, where 0 = not at all confident to 10 = very confident
Fugl Meyer Sensory Evaluation | Baseline, 3 weeks post-intervention and three-months follow-up
  Upper limb sensory function measure with a minimum score of 0 and a maximum score of 12 per domain. A higher score indicates a better somatosensory outcome.
Montreal Cognitive Assessment (MOCA) | Baseline, 3 weeks post-intervention and three-months follow-up
  Cognitive impairment measure. The MoCA is scored out of 30 points. A score below 26 may indicate cognitive impairment.
Upper limb strength | Baseline, 3 weeks post-intervention and three-months follow-up
  Dynamometry measure measuring pincer and power grip force.
Electroencephalography | Baseline and 3 weeks post-intervention
  Cortico-cortical connectivity at rest and ascending somatosensory tract integrity evoked potential measures.
Transcranial magnetic stimulation | Baseline and 3 weeks post-intervention
  Corticospinal tract integrity measures involving motor evoked potential recruitment curves of extensor carpi radialis and first dorsal interosseous muscles.
Magnetic Resonance Imaging (3T) | Baseline
  Volumetric structural MRI including full lesion volume.
Kinematic measures- KINARM | Baseline, 3 weeks post-intervention and three-months follow-up
  Kinematic parameter: 2D reaching (assessed using standardised KINARM tasks with scores below 1.96 considered to be within the normal range)
Kinematic measures- KINETIKOS | Baseline, 3 weeks post-intervention and three-months follow-up
  Kinematic parameter: 3D reaching (assessed using standardised KINETIKOS scapulae movement task which measures the amount movement variability of the scapulae during an arm lift).
Finger individuation | Baseline, 3 weeks post-intervention and three-months follow-up
  The ability to move fingers independently will be assessed using a customised task and an ergonomic device (Hummingbird, Mindmaze) that will independently measure finger strength and dexterity from all digits, in both flexion and extension movements. The device will obtain maximum voluntary force for each finger, and finger individuation, by measuring how much the non-instructed fingers participate when only one instructed finger needs to be moved independently

CONTACTS AND LOCATIONS:
Overall Officials: Nick Ward, MD, Principal Investigator — University College, London
Locations (1):
- Nick Ward, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following the study, access to anonymised data will be strongly regulated and permissions to access the data will be treated on a case-by-case basis.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after primary publication is complete.
Access Criteria: Following the study, access to anonymised data will be strongly regulated and permissions to access the data will be treated on a case-by-case basis.

REFERENCES:
- [Derived] Tedesco Triccas L, Sporn S, Coll I Omana M, Brander F, Kelly K, Bestmann S, Ward N. High-dose high-intensity Queen Square upper-limb rehabilitation for people with chronic stroke (INTENSIVE): protocol for a single-centre, randomised controlled trial. BMJ Open. 2025 Feb 18;15(2):e095766. doi: 10.1136/bmjopen-2024-095766. PMID 39965939